CLINICAL TRIAL: NCT00746668
Title: A Multi-Center Study of Reading Rehabilitation in Macular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: C6246-R
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Age Related Maculopathy; Retinal Degeneration
Keywords: Reading; Macular Degeneration; Rehabilitation; Vision, Low
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration; Vision, Low

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Control Group (Experimental): Subjects randomly assigned to this group had their training delayed for 18 weeks. These subjects underwent four assessments: baseline and at three 6-week intervals' but, they were not given any training during this time. After this data collection period, these control subjects were given training on the three modules. However, their performance after each period of training was not assessed.
  Interventions: Behavioral: Module 1: Visual Awareness and Eccentric Viewing; Behavioral: Module 2: Control of Reading Eye Movements; Behavioral: Module 3: Reading Practice with RSVP
- Group 1 (Experimental): The subjects were trained in 6 weekly sessions of approximately 2 hours each, plus time for rest. This was followed by second assessments. The subjects were then trained on a second module for another 6 weeks, followed by third assessments. Finally, the subjects were trained on a third module for 6 weeks, followed by final assessments.
  Subjects in this group were trained according to the following counterbalanced module order:
  Training Session 1: Module 1 (Visual Awareness and Eccentric Viewing) Training Session 2: Module 2 (Control of Reading Eye Movements) Training Session 3: Module 3 (Reading Practice with RSVP)
  Interventions: Behavioral: Module 1: Visual Awareness and Eccentric Viewing; Behavioral: Module 2: Control of Reading Eye Movements; Behavioral: Module 3: Reading Practice with RSVP
- Group 2 (Experimental): The subjects were trained in 6 weekly sessions of approximately 2 hours each, plus time for rest. This was followed by second assessments. The subjects were then trained on a second module for another 6 weeks, followed by third assessments. Finally, the subjects were trained on a third module for 6 weeks, followed by final assessments.
  Subjects in this group were trained according to the following counterbalanced module order:
  Training Session 1: Module 2 (Control of Reading Eye Movements) Training Session 2: Module 3 (Reading Practice with RSVP) Training Session 3: Module 1 (Visual Awareness and Eccentric Viewing)
  Interventions: Behavioral: Module 1: Visual Awareness and Eccentric Viewing; Behavioral: Module 2: Control of Reading Eye Movements; Behavioral: Module 3: Reading Practice with RSVP
- Group 3 (Experimental): The subjects were trained in 6 weekly sessions of approximately 2 hours each, plus time for rest. This was followed by second assessments. The subjects were then trained on a second module for another 6 weeks, followed by third assessments. Finally, the subjects were trained on a third module for 6 weeks, followed by final assessments.
  Subjects in this group were trained according to the following counterbalanced module order:
  Training Session 1: Module 3 (Reading Practice with RSVP) Training Session 2: Module 1 (Visual Awareness and Eccentric Viewing) Training Session 3: Module 2 (Control of Reading Eye Movements)
  Interventions: Behavioral: Module 1: Visual Awareness and Eccentric Viewing; Behavioral: Module 2: Control of Reading Eye Movements; Behavioral: Module 3: Reading Practice with RSVP
- Group 4 (Experimental): The subjects were trained in 6 weekly sessions of approximately 2 hours each, plus time for rest. This was followed by second assessments. The subjects were then trained on a second module for another 6 weeks, followed by third assessments. Finally, the subjects were trained on a third module for 6 weeks, followed by final assessments.
  Subjects in this group were trained according to the following counterbalanced module order:
  Training Session 1: Module 1 (Visual Awareness and Eccentric Viewing) Training Session 2: Module 3 (Reading Practice with RSVP) Training Session 3: Module 2 (Control of Reading Eye Movements)
  Interventions: Behavioral: Module 1: Visual Awareness and Eccentric Viewing; Behavioral: Module 2: Control of Reading Eye Movements; Behavioral: Module 3: Reading Practice with RSVP
- Group 5 (Experimental): The subjects were trained in 6 weekly sessions of approximately 2 hours each, plus time for rest. This was followed by second assessments. The subjects were then trained on a second module for another 6 weeks, followed by third assessments. Finally, the subjects were trained on a third module for 6 weeks, followed by final assessments.
  Subjects in this group were trained according to the following counterbalanced module order:
  Training Session 1: Module 2 (Control of Reading Eye Movements) Training Session 2: Module 1 (Visual Awareness and Eccentric Viewing) Training Session 3: Module 3 (Reading Practice with RSVP)
  Interventions: Behavioral: Module 1: Visual Awareness and Eccentric Viewing; Behavioral: Module 2: Control of Reading Eye Movements; Behavioral: Module 3: Reading Practice with RSVP
- Group 6 (Experimental): The subjects were trained in 6 weekly sessions of approximately 2 hours each, plus time for rest. This was followed by second assessments. The subjects were then trained on a second module for another 6 weeks, followed by third assessments. Finally, the subjects were trained on a third module for 6 weeks, followed by final assessments.
  Subjects in this group were trained according to the following counterbalanced module order:
  Training Session 1: Module 3 (Reading Practice with RSVP) Training Session 2: Module 2 (Control of Reading Eye Movements) Training Session 3: Module 1 (Visual Awareness and Eccentric Viewing)
  Interventions: Behavioral: Module 1: Visual Awareness and Eccentric Viewing; Behavioral: Module 2: Control of Reading Eye Movements; Behavioral: Module 3: Reading Practice with RSVP

INTERVENTIONS:
Behavioral: Module 1: Visual Awareness and Eccentric Viewing — In this module, awareness of the PRL location and eccentric viewing were trained. Exercises based on published sources were administered. One example of these exercises is the clock face display adapted from Holcomb and Goodrich and Maplesden.
  This module also focused on awareness of the perceptual consequences of using a PRL. The purpose of these training exercises was to allow the subjects to appreciate perceptual alterations that occur when using a PRL and to practice making perceptual discriminations with the peripheral retina. Previously published work has demonstrated that perception in the peripheral retina can be affected by practice.
Behavioral: Module 2: Control of Reading Eye Movements — In this module, control of eye movements was trained. These exercises began with a series of saccade tasks to nonalphabetical stimuli and then progressed to single letter, letter pairs, and word stimuli. Subjects were instructed to make a saccade between the dots. The experimenter provided feedback concerning the appropriateness of the saccades, and the alternation rate of the dots was increased as performance improved.
Behavioral: Module 3: Reading Practice with RSVP — In module 3, we wanted to assess only the higher-level effects of reading practice. Subjects practiced reading using stimuli that did not require reading eye movements. An example is short sentences that were presented one word at a time at a single location on a screen (Rapid Serial Visual Presentation [RSVP]). At the end of the sentence, subjects reported whether the sentence made sense or not. We also had our subjects practice reading scrolled text. Although, eye movements and saccades may spontaneously occur under the text presentation conditions of this module, they are not the efficient saccades necessary for reading.
  Other Names: Sequential Presentation of Lexical Information

SUMMARY:
The purpose of this study is to measure the effectiveness of a newly-designed oculomotor training program for patients with macular disease, including age-related macular degeneration.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is currently among the top three leading causes of central vision loss in veterans (Chomsky et al., 1995) and is the most prevalent cause of blindness among veterans (37.2%, Quillen & Henry, 2000). The loss of central vision associated with these diseases has a profound impact on the quality of life to those affected, with many suffering depression. It is devastating to no longer be able to read a newspaper or recognize facial expressions. The use of preferred retinal locations (PRLs) to compensate for diseased foveae has offered hope to these patients in regaining some function. The investigators have developed a protocol that includes training in two major visual skills areas:

* Visual awareness and eccentric viewing; and
* Reading practice with sequentially lexical information

Module 1 focuses on making the patient aware of better vision at an eccentric location relative to degraded vision at the diseased fovea. Module 2 is focused on reading practice without eye movements. These program curriculums and preliminary results are provided in the present proposal. The primary aim of this proposal is to quantitatively assess the relative effectiveness for improving reading and to establish the minimum training time need for skill improvement. One hundred and twenty patients with macular disease who are already using a PRL and similar in visual characteristics (e.g., visual acuity, contrast sensitivity, size of scotoma, duration of the disease) will be included the study. All patients will be trained with both modules using a repeated measures-completely counterbalanced - design to control for training order effects. In addition, all patients will be assessed using the same outcome measures of reading (using MNRead Acuity Charts and the View Sentences Test). The performance of the patients on the outcomes battery post-training will be compared to their pre-training performance on the same battery. Questionnaires (the Veterans Administration Low Vision Visual Functioning Questionnaire, CES-D, Short Form-36, and Adaptation to Vision Loss Scale) will also be administered to assess perceived abilities to perform everyday tasks, adaptation to vision loss, moods, and general health. In addition, patients will also be assessed on the exercises practiced during the module at the end of each daily training session to determine exactly when in the training protocol an improvement in performance on the exercises being trained has occurred. These daily performance measures provide for a finer scale for detecting performance changes. Statistical analyses will be conducted to answer the following questions:

* Does a combination of eccentric viewing awareness and oculomotor training produce significant improvements in reading rate?
* Which exercises are most effective in training the visual skills associated with reading and at what point during the course of training do the patients reach asymptotic performance?
* How do co-factors such as age, PRL size and location, and cognitive capabilities relate to training outcomes?

Advancements are being made in the area of retinal cell transplantation, gene therapy, and retinal prosthetics. When these techniques become part of the standard clinical care, it is likely that all the patients will require vision rehabilitation techniques to help them make sense of their potentially fragmented percepts. This research offers an evaluation of relative successes of the components of reading rehabilitation and will lead to the design of an efficient and effective composite training strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of macular disease, such as age-related macular degeneration
* An established preferred retinal locus
* Visual acuity of less than or equal to 20/70 and greater than or equal to 20/400 (in the better eye)

Exclusion Criteria:

* Those with other major ophthalmologic and neurologic disease
* choroidal neovascularization ("wet" AMD)
* moderate to severe media opacities, and cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet P Szlyk, PhD, Principal Investigator — Jesse Brown VAMC (WestSide Division)
Locations (1):
- Jesse Brown VAMC (WestSide Division), Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Started | 6 | 5 | 5 | 5 | 5 | 5 | 5
Completed | 6 | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All subjects' reading performances were initially assessed before training began. Reading performance were assessed using sentences displayed on a computer monitor. Two lines of text were presented at the center of the monitor with each subject seated at a viewing distance of 40cm. The subject read each sentence aloud and indicated whether it made sense by responding true or false. Reading speed was calculated using an algorithm similar to that used for the MNRead test.
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Sentence Reading
Description: To assess reading performance, after each training module (1-3), two lines of text were presented at the center of the monitor. Each subject was seated with his or her forehead on a head rest at a viewing distance of 40cm. The subject read each sentence aloud and indicated whether it made sense by responding true or false. Reading speed was calculated using an algorithm similar to that used for the MNRead test. The number of words read correctly was divided by the time required to read the sentence to yield a measure of reading speed in words per minute (wpm). Sentences were displayed at sizes of 0.1, 0.2, 0.3, 0.4, 0.5, and 0.6 log units above the subject's letter acuity threshold. Five sentences were presented at each font size. We used 105 different sentences so that no sentence was repeated for any subject. Average speed of reading (log wpm) was plotted as a function of font size (logMAR).
Time Frame: Pre-training, 6 weeks, 12 weeks, 18 weeks
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Words per Minute (wpm)
Groups:
- Arm 1: Pre-Training: Baseline Assessment prior to training.
- Arm 2: Assessment After Module 1: Assessment after six-weeks of training in Module 1 (PRL Awareness Training).
- Arm 3: Assessment After Module 2: Assessment after six-weeks of training in Module 2 (Eye Movement Training).
- Arm 4: Assessment After Module 3: Assessment after six-weeks of training in Module 3 (RSVP Reading).
Arm/Group | Arm 1: Pre-Training | Arm 2: Assessment After Module 1 | Arm 3: Assessment After Module 2 | Arm 4: Assessment After Module 3
Number analyzed (Participants) | 30 | 30 | 30 | 30
Words per Minute (wpm) | 58.9 (0.00) | 50.5 (7.2) | 86.2 (6.8) | 49.1 (7.2)

ADVERSE EVENTS:
Groups:
- Group 1: The subjects were trained in 6 weekly sessions of approximately 2 hours each, plus time for rest. This was followed by second assessments. The subjects were then trained on a second module for another 6 weeks, followed by third assessments. Finally, the subjects were trained on a third module for 6 weeks, followed by final assessments.
  Subjects in this group were trained according to the following counterbalanced module order:
  Training Session 1: Module 1 (Visual Awareness and Eccentric Viewing) Training Session 2: Module 2 (Control of Reading Eye Movements) Training Session 3: Module 3 (Reading Practice with RSVP)
  .
Arm/Group | Control Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes